CLINICAL TRIAL: NCT00585793
Title: Study of the Relationship Between HIV-1 Subtype and Antiretroviral (ARV) Response in Ugandan Children
Brief Title: Relationship Between HIV-1 Subtype and ARV Response
Acronym: RELATES
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: H-2006-0206
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: HIV Infections
Keywords: HIV/AIDS
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — lopinavir-ritonavir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma obtained from participants
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PEPFAR 1
  Interventions: Drug: NRTI/NNRTI/ Kaletra

INTERVENTIONS:
Drug: NRTI/NNRTI/ Kaletra — Fixed dose and cild formulation Kaletra

SUMMARY:
Does subtype of HIV-1 affect the response of ARVs given to Ugandan children

DETAILED DESCRIPTION:
There is a growing demand for treatment and access to antiretroviral (ARV) therapy for HIV infection in resource - poor settings. Of all the HIV-1 subtypes (A, B, C, D, F, G, H, J, K and multiple recombinant viruses), ARV drugs were developed by studying primarily subtype B. This HIV subtype predominates in North America, Western Europe and the rest of the industrialized world. However, worldwide, subtype B makes up a minority (about 10%) of the HIV infected population. In Uganda, HIV-1 subtypes A and D predominate. Although there is some evidence that the ARV's developed against subtype B virus have activity against non-subtype B virus, as the demand grows for ARV's in resource-poor settings, it is not entirely clear whether all non-B subtypes will respond robustly to the current ARV's available. Also, it is unknown if drug failure (in the form of viral resistance) to non-subtype B virus is due to mutations that are similar to those seen in subtype B virus. Without more data in resource-poor countries, it is still too early to tell whether different HIV-1 subtypes will require unique drug treatment or salvage strategies for those who fail initial therapy.

The University of Wisconsin (UW) Health HIV Care Program has been partnering with the Mulago Hospital Pediactirc Infectious Disease Clinic (PIDC) for the past five years. The PIDC has well over 5,000 children with HIV that attend this clinic. Approximately 20% of these children have met criteria for ARV treatment under the US PEPFAR (Presidents Emergency Plan for AIDS Relief) arrangement. A retrospective collaborative (UW/PIDC) study performed at the PIDC examined (using genotyping) 40 children who failed initial ARV therapy. This study found some different mutations in children who failed the antiretroviral therapy.

Based upon the above study, the goal of the present cohort study is to examine prospectively in an expanded population of children who attend the PIDC the relationship between the HIV subtype infecting Ugandan children and their virologic and clinical response to the ARV's now available to this population. Approximately 30% of children are currently failing (based primarily upon clinical data) ARV therapy at the PIDC. In this study, these children will have a separate tube of 5 cc of blood drawn (at specified times) for HIV subtyping to examine whether specific subtypes of HIV are associated with failure to specific ARV's or ARV combinations. In addition to HIV subtype determination, viral genotyping (viral mutations) will be performed to examine the relationship between the HIV subtype and specific viral mutations indicating resistance to an ARV.

The overall design of this study is to prospectively collect cohort clinical and virologic data from children (ages birth to 16 years) started on ARV therapy during a 12 month period of enrollment (about 110 children who qualify for PEPFAR ARV treatment). The only inclusion criteria is the child receives ARV therapy. The only exclusion is refusal on the part of the patient or family to have blood drawn and records examined. Children receiving ARV therapy in this time period will be approached and recruited for this study by the attending physician. This study is approved by the University of Wisconsin Hospital and Clinics and Mulago Hospital IRBs.

All treated children will have clinical and HIV genotype and subtype data (blood sent to U. Wisconsin for analysis) collected prior to starting ARV's. Children will then receive as initial therapy for HIV infection 2 NRTIs (AZT, d4T, ABC or ddI) and 1 NNRTI (Neverapine, or Efavirenz) or Kaletra (a protease inhibitor). One month after starting ARVs (and every four months thereafter during the study period) an HIV viral load will be obtained. If the child is failing therapy, clinical data at the time of failure will be collected and blood will be drawn for repeat viral load, HIV-1 subtyping (has the subtype changed), and genotypic analysis (see below). Decisions on what to use as treatment for those children failing their first antiretroviral regimen will be made using the data collected on the blood obtained from each child in the study.

ARV failure at the PIDC is generally assessed on clinical grounds (weight loss, diarrhea, fever, opportunistic infection [OI] etc). The PIDC has a fairly sophisticated data management system. In those children having clinical failure to the ARV's after initial therapy, blood for HIV-1 viral load, subtype and genotype will be drawn. This blood will be frozen and shipped to the University of Wisconsin for analysis. On site (Dr. Kekitiinwa) clinical data will be collected. This data will include age, sex, physical findings and clinical course on ARV's. More specifically, the reason for ARV failure was: the occurrence of OI, wasting, recurrence of diarrhea, (other symptoms of HIV), or toxicity to the ARV (tolerability). All blood samples will be labeled only with a number that corresponds to the identity of the patient. This number will be kept by Dr. Graziano. These samples will then be Federal Expressed on dry ice to the University of Wisconsin where they will be evaluated for HIV-1 subtype and genotype.

No material inducements for recruitment will be offered and no personnel at the PIDC will receive incentives for recruitment of subjects.

This study is minimal risk to the patient. ARV therapy is standard of care at the PIDC for those infected with HIV and having AIDS.

T-tests of significance and other population cohort analyses will be performed to examine whether there is a correlation between HIV-1 subtype, clinical failure, and the appearance of specific genetic resistant mutants. There is no statistical justification for the sample size.

The only risk from this study is bruising and the transient pain of the blood drawn for analysis (see consent form). Since AIDS is a devastating disease in Uganda and ARV therapy represents the only hope HIV infected children have, there is no particular concern for examination of medical records for these children. There is no cultural sensitivity to drawing blood in PIDC population.

The clinical benefit to the study participants in this research is the knowledge of mutations (in those failing therapy) before starting second line therapy.

Physicians caring for the patient will administer the consent form. All are fluent in English (the national Uganda language) and Lugandan (the prevalent dialect in Kampala and surrounding areas). See the consent form (What your signatures or thumb print means) enclosed for details.

FMG:misc/Study Description.doc

ELIGIBILITY:
Inclusion Criteria:

* PEPFAR eligible

Exclusion Criteria:

* OI/sfaety lab abnomalities

Ages: 4 Months to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children $ ,monthe to 16 years
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2008-07; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
HIV-1 subtype affects response to ARVs | 3 years

SECONDARY OUTCOMES:
Comparison of NNRTI/NRTI combinations to Kaletra/NRTI combinations in Ugandan Children | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Frank M Graziano, MD/PhD, Principal Investigator — UWHC
Locations (1):
- Kampala, Uganda